CLINICAL TRIAL: NCT01017484
Title: Mechanism of the Blood Pressure Lowering Effect of the DASH Dietary Pattern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Pro00001236; AHA 0755460U (Other: AHA)
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2009-11

CONDITIONS: Blood Pressure
Keywords: blood pressure; DASH diet; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DASH (Experimental): The Dietary Approaches to Stop Hypertension Dietary pattern.
  Interventions: Other: DASH, Control
- Control (Experimental): The typical American diet as estimated from the NHANES survey.
  Interventions: Other: DASH, Control

INTERVENTIONS:
Other: DASH, Control — controlled feeding of either the DASH dietary pattern or a typical American diet at isocaloric level.

SUMMARY:
Understanding the possible mechanism(s) by which the DASH dietary pattern lowers blood pressure will potentially enhance the value of this dietary intervention by elucidating the conditions under which it will be most effective, identifying target populations, examining its impact on vascular health beyond blood pressure, and enhancing the investigators' understanding of the interactions among diet, blood pressure and vascular function. In addition, results of this study may help to identify additional therapeutic targets. Therefore, the overall goal of the proposed study is to determine the mechanism(s) by which the DASH dietary pattern lowers blood pressure by using a controlled feeding design.

DETAILED DESCRIPTION:
Randomized, controlled feeding trials have established the BP lowering effects of the Dietary Approaches to Stop Hypertension (DASH) dietary pattern, which emphasizes fruits, vegetables and low fat dairy and is low in saturated and total fat. The DASH studies were designed to establish efficacy, not to determine mechanism of action. Other studies suggest that the DASH diet may have effects on the renin-angiotensin-aldosterone system (RAAS). These effects have not been directly evaluated, nor have other potential mechanisms of action such as effects on adrenergic tone, vascular function and inflammation. The BP-lowering effect of the DASH dietary pattern was maximal after two weeks of controlled feeding, and was comparable in magnitude to antihypertensive medication among participants with stage 1 hypertension. Understanding the possible mechanism(s) by which the DASH diet lowers BP will potentially enhance the value of this intervention by elucidating the conditions under which it will be most effective, identifying target populations, examining its impact on vascular health beyond BP, and enhancing our understanding of the interactions among diet, BP and vascular function. In addition, results of this study may help to identify additional therapeutic targets. Therefore, the overall goal of the proposed study is to determine the mechanism(s) by which the DASH diet lowers BP. Our unifying hypothesis is that DASH diet lowers BP through effects on vascular function and sodium excretion, mediated through the effects on RAAS.

ELIGIBILITY:
Inclusion Criteria:

1. SBP 140-159 mm Hg and DBP 90-99 mm Hg based on mean values over two screening visits,
2. Age ≥22 years, and
3. Willing to eat at least one on-site meal/day, five days/week, and willing to eat study diets and nothing else for the 3 weeks of controlled feeding.

Exclusion Criteria:

1. Any serious illness that would interfere with participation or make DASH diet unsafe to the participants,
2. Currently on cancer chemotherapy or with evidence of active malignancy or radiation therapy within past six months,
3. History of CVD event (MI, CABG, angioplasty, symptomatic ischemic heart disease, or stroke),
4. Clinical diagnosis of congestive heart failure,
5. Current diagnosis of diabetes and treatment for diabetes with oral medication or insulin,
6. Body mass index > 45 Kg/m2,
7. DASH MECHANISM staff or household member of DASH MECHANISM staff,
8. Using Medications including BP lowering drugs within the last three months, using lithium,insulin or oral diabetes medications, oral corticosteroids, unstable doses of psychotropics or phenothiazines, antacids or nutritional supplements unless they can be discontinued, or weight reducing medications;
9. Consumption of more than 14 alcoholic drinks per week;
10. Investigator discretion for safety or compliance reasons;
11. Inability to provide reliable BP & vascular functions measurements;
12. Planning to leave the area prior to the anticipated end of the intervention period;
13. Pregnant, planning a pregnancy prior to the end of intervention, or breast feeding;
14. Significant food allergies, preferences, or dietary requirements that would interfere with diet adherence; and
15. Subjects taking medications for erectile dysfunction.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
urinary sodium | 2 weeks

SECONDARY OUTCOMES:
blood pressure | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Hwa Lin, PhD, Principal Investigator — Duke University